CLINICAL TRIAL: NCT05952180
Title: Effect of Virtual Reality Combined With Cycloergometer Versus Conventional Cycloergometer on Distance for ICU Non-sedated Participants: Prospective Randomized Controlled Trial
Brief Title: Effect of Virtual Reality Combined With Cycloergometer Versus Conventional Cycloergometer on Distance Covered for Intensive Care Unit Non-sedated Participants
Acronym: CYCLOREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2023-03
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Intensive Care Unit
Keywords: Virtual Reality exercise; Early Rehabilitation; Intensive care unit; lower limb/upper limb; Postoperative Period; cycloergometer

STUDY DESIGN:
Intervention Model Description: Monocentric cross-over trial comparing the combination of cycloergometer and virtual reality to standard cycloergometer, in ICU, over the actively covered distance in kilometers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality and Cycloergometer (Experimental): The session performed uses a standard cycloergometer, with the participant pedaling in a seated position with the lower limbs. A 43 inches TV screen is placed in front of the cycloergometer where the participant will watch a video of a walk through a natural environment on. The speed of the walk is linked to the pedaling speed so that the faster the participant pedals, the faster the video goes too. The session last 30 minutes in the participant's room.
  Interventions: Device: Virtual reality and Cycloergometer
- Standard cycloergometer (Active Comparator): For the "standard cycloergometer" intervention, the session uses usual cycloergometer with the participant pedaling in a seated position with the lower limbs. No virtual reality is used. The session last 30 minutes in the participant's room
  Interventions: Other: Standard cycloergometer

INTERVENTIONS:
Device: Virtual reality and Cycloergometer — The session performed uses a standard cycloergometer, with the participant pedaling in a seated position with the lower limbs. A 43 inches TV screen is placed in front of the cycloergometer where the participant will watch a video of a walk through a natural environment on. The speed of the walk is linked to the pedaling speed so that the faster the participant pedals, the faster the video goes too. The session last 30 minutes in the participant's room.
  Arms: Virtual reality and Cycloergometer
Other: Standard cycloergometer — the session uses usual cycloergometer with the participant pedaling in a seated position with the lower limbs. The session lats 30 minutes in the participant's room.
  Arms: Standard cycloergometer

SUMMARY:
Management in intensive care unit (ICU) has gradually evolved to early mobilization. Studies have confirmed a 50% decrease impact on the functional abilities and quality of life after ICU. The cycloergometer is particularly studied and effective for early rehabilitation. Current practices encounter obstacles as fatigue, pain or a lack of motivation to mobilize. Several studies have been carried out to evaluate the effects of virtual reality (VR) on mental health and on cognitive abilities. To date, there is little evidence about VR on distraction and the impact on physical activity motivation in ICU.

The main hypothesis is that the use of combine cycloergometer and VR would improve the travelled distance by patients in ICU. Adverse effects would be observed initially in order to consolidate the safety data of this device. It would also allow a better participant experience.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old hospitalized in the surgical intensive care unit (USC or reanimation) of the Centre Hospitalier Régional d'Orléans
* Glasgow 15
* Satisfying the chair installation criteria before the inclusion
* With or without :

  * any type of invasive or non-invasive ventilation
  * any type of oxygenation
* Stable within its medically determined target parameters
* Hemodynamically stable (MAP>65)

Exclusion Criteria:

* Person presenting a medical contraindication to cycloergometer
* Person under guardianship or curatorship
* Person under court protection
* Stay less than 48 hours (post-neurosurgery surveillance)
* Persons weighing over 180 kg
* Person not affiliated to a social security system
* Pregnant or breast-feeding Women
* Deaf and visually impaired people
* Patient included in another study with the same endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Distance actively covered (in kilometers with one decimal) | Day 2
  Distance actively covered (in kilometers) with the combination of virtual reality and cycloergometer versus distance actively covered (in kilometers with one decimal) with conventional seated cycloergometer session

SECONDARY OUTCOMES:
Number of adverse effects noted during the session | Day 2
  Compare between the two cross-over groups the adverse effects noted during the session
Measure of patient's experience with Visual Analogic Scale (on /10) | Day 2
  Compare between the two cross-over groups - the patient's experience of "perception of effort", "sensation of escape from the virtual reality" and "motivation to a next session"

CONTACTS AND LOCATIONS:
Locations (1):
- CHR d'Orléans, Orléans, France

REFERENCES:
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Nickels MR, Aitken LM, Barnett AG, Walsham J, McPhail SM. Acceptability, safety, and feasibility of in-bed cycling with critically ill patients. Aust Crit Care. 2020 May;33(3):236-243. doi: 10.1016/j.aucc.2020.02.007. Epub 2020 Apr 18. PMID 32317212
- [Background] Dubb R, Nydahl P, Hermes C, Schwabbauer N, Toonstra A, Parker AM, Kaltwasser A, Needham DM. Barriers and Strategies for Early Mobilization of Patients in Intensive Care Units. Ann Am Thorac Soc. 2016 May;13(5):724-30. doi: 10.1513/AnnalsATS.201509-586CME. PMID 27144796
- [Background] Wada T, Matsumoto K, Arai M. [Nursing of patients with diseases of digestive or endocrine organs]. Kurinikaru Sutadi. 1988 Nov;9(12):1174-9. No abstract available. Japanese. PMID 3210786
- [Background] Warburton DE, Bredin SS, Horita LT, Zbogar D, Scott JM, Esch BT, Rhodes RE. The health benefits of interactive video game exercise. Appl Physiol Nutr Metab. 2007 Aug;32(4):655-63. doi: 10.1139/H07-038. PMID 17622279
- [Background] Monedero J, Lyons EJ, O'Gorman DJ. Interactive video game cycling leads to higher energy expenditure and is more enjoyable than conventional exercise in adults. PLoS One. 2015 Mar 4;10(3):e0118470. doi: 10.1371/journal.pone.0118470. eCollection 2015. PMID 25738290